CLINICAL TRIAL: NCT05504798
Title: Efficacy of Neuromuscular Electrical Stimulation and Interrupted Serial Casting in Children With Spastic Diplegic Cerebral Palsy
Brief Title: A New Multimodal Treatment Approach for Children With Spastic Diplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasser Mamdouh Abd Elmonem Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003675
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-08

CONDITIONS: Spastic Diplegic Cerebral Palsy
Keywords: Diplegia, Neuromuscular electrical stimulation, Casting.
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Active Comparator): will receive a selected physical therapy program.
  Interventions: Other: Selected physical therapy program
- Group (B) (Active Comparator): will receive interrupted progressive serial casting in addition to a modified selected physical therapy program during casting.
  Interventions: Other: Selected physical therapy program; Procedure: Interrupted serial casting
- Group (C) (Active Comparator): will receive interrupted progressive serial casting and the modified selected physical therapy as group (B) in addition to neuromuscular electrical stimulation for ankle dorsiflexors and knee extensors muscles through cast windows
  Interventions: Other: Selected physical therapy program; Procedure: Interrupted serial casting; Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Selected physical therapy program — Selected physical therapy program one hour three times weekly for six successive weeks including stretching, strengthening, balance, and gait training.
Procedure: Interrupted serial casting — Interrupted casting for 5 days a week for six successive weeks using a dual cast which consists of a standard short leg cast and a circular cast from below the knee to above the knee.
  Arms: Group (B); Group (C)
Device: Neuromuscular electrical stimulation — Neuromuscular electrical stimulation in form of faradic current with frequency of 50 Hz, and intensity of maximum tolerable intensity to produce a visible contraction but as tolerated by the child for ankle dorsiflexors and knee extensors muscles through cast windows over the motor points of these muscles for 30 min 3 times weekly for six successive weeks
  Arms: Group (C)

SUMMARY:
Combining the advantages of both Neuromuscular electrical stimulation and lower limb serial casting to a selected physical therapy program in children with spastic diplegic cerebral palsy to overcome the adverse effects during the period of casting and the long period of rehabilitative interventions, providing a new multimodal treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* The children will have grade 2 or 3 on Modified Ashworth Scale.
* The children will have Level II, or III according to the Gross Motor Function Classification System.
* The children walk with equinus or jump gait patterns with spasticity of the hamstrings and hip flexors in addition to calf muscles spasticity.
* Children take their Antispastic drug use such as baclofen, diazepam or tizanidine.
* All children will be able to follow instructions.

Exclusion Criteria:

* children will be excluded from the study if they have any problems of the following:

  * Cognitive dysfunction.
  * Poor skin integrity.
  * History of or recent nonunion fracture.
  * Fixed contractures and deformities.
  * Previous surgery (tendon lengthening).
  * Received Botulinum toxin A injections in the last six months.
  * Impaired circulation.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of knee and ankle passive range of motion (ROM) | At the beginning and after six weeks of intervention
  Digital Goniometer will be used to measure the passive ROM of ankle dorsiflexion and the popliteal angle (PA)
Change of strength of knee extensors and ankle dorsiflexors muscles | At the beginning and after six weeks of intervention
  Hand-held dynamometers (HHDs) " Lafayette manual muscle tester" (MMT) Will be used for quantitative assessment of maximal voluntary isometric contraction for knee extensors, and ankle dorsiflexors.
Change of tone of hamstring and gastrocnemius muscles | At the beginning and after six weeks of intervention
  The Modified Tardieu Scale (MTS) will be used for analysis of dynamic spasticity of gastrocnemius and hamstring muscles. Measuring R1 (the fast velocity movement of the ankle or knee through the full ROM to determine the point of catch in the ROM), R2 (the passive ROM), and R2-R1 (dynamic component of spasticity).

SECONDARY OUTCOMES:
Change in sagittal kinematics parameters of gait pattern | At the beginning and after six weeks of intervention
  The Observational Gait Scale (OGS) will be used for analysis of gait kinematics through 2 D videography with slow motion and split-screen video. Six sections will be tested to evaluate knee and ankle kinematics (Knee position in mid stance, Initial foot contact, Foot contact at mid stance, Base of support, Gait assistive devices, degree of change) with a total score of 17 on each limb. the minimum score is -2 and maximum score is 17. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No